CLINICAL TRIAL: NCT06936527
Title: An Open-label, Multicenter Phase Ib/II Clinical Study: Aim to Valuate the Efficacy and Safety of XS-03 Comination With FOLFOX or FOLFIRI and Bevacizumab in Metastatic Colorectal Cancer Patients With RAS Mutation
Brief Title: XS-03 in Combination With FOLFOX or FOLFIRI and Bevacizumab for Treatment of Metastatic Colorectal Cancer Patients With RAS Mutation
Acronym: XS-03-II201
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NovaOnco Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XS-03-II201
Record Dates: First submitted 2025-04-02; First posted 2025-04-20 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer; Metastatic Colorectal Cancer With RAS Mutation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental arm 1: XS-03 + FOLFOX/FOLFIRI + Bevacizumab (Experimental): Phase 1b: XS-03 escalating orally Day 1 through Day 5 and Day 15 through Day 19 of each 28-day cycle in combination with FOLFOX or FOLFIRI and bevacizumab.
  FOLFOX (85 mg/m^2 oxaliplatin, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-fluorouracil (5-FU), and 2400 mg/m^2 continuous intravenous infusion 5-FU) , 5 mg/kg bevacizumab FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-fluorouracil (5-FU), and 2400 mg/m^2 continuous intravenous infusion 5-FU), 5 mg/kg bevacizumab
  Interventions: Biological: Drug: XS-03, Biological: Bevacizumab, Drug: FOLFOX, Drug: FOLFIRI
- Experimental arm 2: XS-03 + FOLFOX/FOLFIRI + Bevacizumab (Experimental): Phase 2: XS-03 Recommended Phase 2 Dose (RP2D) and selected one more dosage orally Day 1 through Day 5 and Day 15 through Day 19 of each 28-day cycle in combinationwith FOLFOX or FOLFIRI and bevacizumab.
  FOLFOX (85 mg/m^2 oxaliplatin, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-fluorouracil (5-FU), and 2400 mg/m^2 continuous intravenous infusion 5-FU) , 5 mg/kg bevacizumab FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-fluorouracil (5-FU), and 2400 mg/m^2 continuous intravenous infusion 5-FU), 5 mg/kg bevacizumab
  Interventions: Biological: Drug: XS-03
- Comparator: FOLFOX/FOLFIRI + Bevacizumab (Active Comparator): Phase 2: Comparator arm treat with FOLFOX or FOLFIRI + bevacizumab intravenously.
  FOLFOX (85 mg/m^2 oxaliplatin, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-fluorouracil (5-FU), and 2400 mg/m^2 continuous intravenous infusion 5-FU) , 5 mg/kg bevacizumab FOLFIRI (180 mg/m^2 irinotecan, 400 mg/m^2 leucovorin, 400 mg/m^2 bolus 5-fluorouracil (5-FU), and 2400 mg/m^2 continuous intravenous infusion 5-FU), 5 mg/kg bevacizumab
  Interventions: Biological: Biological: Bevacizumab, Drug: FOLFOX, Drug: FOLFIRI

INTERVENTIONS:
Biological: Drug: XS-03, Biological: Bevacizumab, Drug: FOLFOX, Drug: FOLFIRI — XS-03 orally Bevacizumab intravenously FOLFOX intravenously FOLFIRI intravenously
  Arms: Experimental arm 1: XS-03 + FOLFOX/FOLFIRI + Bevacizumab
Biological: Drug: XS-03 — XS-03 orally
  Arms: Experimental arm 2: XS-03 + FOLFOX/FOLFIRI + Bevacizumab
Biological: Biological: Bevacizumab, Drug: FOLFOX, Drug: FOLFIRI — Bevacizumab intravenously FOLFOX intravenously FOLFIRI intravenously
  Arms: Comparator: FOLFOX/FOLFIRI + Bevacizumab

SUMMARY:
XS-03 in combination with FOLFOX or FOLFIRI and Bevacizumab for treatment of metastatic colorectal cancer patients with RAS mutation

ELIGIBILITY:
Inclusion Criteria

1. Voluntarily participate in the clinical trial and sign the informed consent form.
2. Age ≥18 and ≤ 70 years. No gender restrictions.
3. Patients with histologically and/or cytologically confirmed metastatic colorectal cancer who are not suitable for surgical treatment.
4. Advanced or metastatic colorectal cancer: Stage Ib patients must have received at least one prior systemic therapy; Stage II patients have no prior systemic therapy. For patients with previously neoadjuvant/adjuvant therapy, disease progression must occur no less than 6 months after the end of therapy to be eligible for inclusion.
5. Documentation of RAS mutation. The previously gene test report issued by qualified testing institution is acceptable. BRAF status is not restricted.
6. Consent to provide tumor tissue samples and peripheral blood for biomarker analysis.
7. Has measurable extracranial lesion according to RECIST v1.1 criteria, defined as at least one lesion that has not received radiotherapy. For previously radiotherapy lesion, there must be imaging evidence of progression after radiotherapy.
8. Eastern Cooperative Oncology Group (ECOG) performance status score 0-1.
9. Expected life expectancy ≥ 6 months.
10. The patient has adequate hepatic, renal and bone marrow function.
11. For a woman of child-bearing potential must have a negative serum pregnancy test within 7 days prior to enrollment. Woman of child-bearing potential and fertile men must agree to use adequate contraception for the duration of study participation and for 6 months after the last dose.

Exclusion Criteria

1. Patients with known high microsatellite instability (MSI-H) or mismatch repair deficiency (dMMR) primary or metastatic colorectal cancer and suitable for immune checkpoint inhibitor treatment assessed by investigators.
2. Previously received bevacizumab and its biosimilar therapy. (Only for phase II)
3. Central nervous system metastases which are symptomatic or require therapy.
4. Imaging shows major blood vessel invasion (such as the aorta, pulmonary artery, pulmonary vein, vena cava, etc.).
5. Adverse events and/or complications that caused by previous antitumor therapy have not recovered to baseline level or ≤ CTCAE grade 1.

   Baseline level or ≤ Grade 1. However, any grade of alopecia, pigmentation, or ≤ Grade 2 peripheral sensory neuropathy, or other conditions assessed by the investigator as having become chronic and not affecting the safety of the study medication are allowed for inclusion.
6. With a history of other malignancies within 5 years or with other malignancies currently prior to screening, except colorectal cancer. Exception: curatively treated early-stage malignancies (in situ carcinoma or stage I tumors), such as adequately treated basal cell or squamous cell skin cancer or in situ cancer of the cervix.
7. Patients have a significant risk of bleeding.
8. Patients have a significant risk of thrombus.
9. Patients have severe cardiovascular disease, including but not limited to: Ischemic heart disease within the past 6 months prior to screening; coronary artery disease post-surgery or stent implantation within 6 months; New York Heart Association (NYHA) functional classification ≥ Class II within 6 months prior to screening; or known left ventricular insufficiency (LVEF <50%)；severe arrhythmia requiring clinical intervention; any other cardiovascular disease that researchers regard the patient unsuitable for participation in the study.
10. Patients with a significantly increased risk of QTc prolongation.
11. Patients unable to swallow drugs or have severe diseases that significantly affect drug absorption.
12. Patients have one of the following viral active infections: active hepatitis B or C; human immunodeficiency virus (HIV) infection; active syphilis
13. During screening, the presence of interstitial lung disease, interstitial pneumonia, pulmonary interstitial fibrosis requiring therapy, or a history of pneumonia caused by tyrosine kinase inhibitors.
14. Patients received radiotherapy within the past 4 weeks prior to the first first dose of study drug.
15. Patients received therapeutic surgeries (excluding diagnosis, biopsy, or drainage procedures) within the past 4 weeks prior to the first dose of study drug, including local treatments such as radiofrequency ablation for liver metastases, or are expected to have major surgeries during the study period.
16. Severity infection need intravenous infusion of antibiotics, antiviral drugs, or hospitalisation within the past 2 weeks prior to the first dose of study drug.
17. Patients must use strong CYP3A4 inducers or inhibitors within the past 2 weeks prior to the first administration, or during the anticipated study period,
18. History of severe allergy, or known allergy to any active or inactive components of the study drug product.
19. Pregnancy or lactation.
20. Patients with severe diseases of any organs or systems, any clinical or laboratory test abnormalities, or other reasons that investigator assess them unsuitable to participate in this clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Number of participants with Dose-limiting Toxicities (DLTs) in experimental arm of XS-03 in combination with FOLFOX or FOLFIRI and Bevacizumab | up to day 28
  Dose-limiting toxicities were defined as events related to XS-03 that were considered an adverse reaction or suspected adverse reaction during the first cycle of treatment
Phase 1b: Determine the Maximum Tolerated Dose (MTD) in experimental arm of XS-03 in combination with FOLFOX or FOLFIRI and Bevacizumab | up to day 28
  MTD is defined as at most 1 patient out of 6 experiencing DLT
Phase 2: Objective Response Rate (ORR) of two experimental arms and comparator arm | up to 18 months after first dose of last patient
  Defined as the percentage of participants that achieve a best overall response of complete response (CR) or partial response (PR) (per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria)

SECONDARY OUTCOMES:
Phase 1b: Objective Response Rate (ORR) of all treated participants | up to 18 months after first dose of last patient
Duration of response (DOR) of all treated participants | up to 18 months after first dose of last patient
  Duration of response defined as time from when response was first documented until first documented disease progression or death, whichever occurs first.
Progression-free survival (PFS) of treated participants | up to 18 months after first dose of last patient
  as determined based on RECIST version 1.1 criteria
Overall survival (OS) of treated participants | up to 18 months after first dose of last patient
  Time in months from date of first dose for phase 1b and randomization for phase 2 to death due to any cause
Number of Participants With Adverse Events (AEs) of treated participants | up to 28 days after last dose of study drug
  The severity of each AE will be graded using the Common Terminology Criteria for Adverse Events (CTCAE).
Number of Participants With Clinically Significant Change From Baseline in safety monitoring | up to 28 days after last dose of study drug
Number of Participants With dose adjustment | up to 28 days after last dose of study drug
  AE associated with dose reduction, interruption and discontinuation
Time to Reach Maximum Peak Plasma Concentration (Tmax) | From pre-dose on day 1 of cycle 1 to day 5 of cycle 3 (28-day cycle length)
  Pharmacokinetic parameter
Maximum Plasma Concentration(Cmax) | From pre-dose on day 1 of cycle 1 to day 5 of cycle 3 (28-day cycle length)
  Pharmacokinetic parameter
Area under the plasma concentration versus time curve from time zero to the last measurable concentration(AUC0-t) | From pre-dose on day 1 of cycle 1 to day 5 of cycle 3 (28-day cycle length)
  Pharmacokinetic parameter
Elimination Half-life (T1/2) | From pre-dose on day 1 of cycle 1 to day 5 of cycle 3 (28-day cycle length)
  Pharmacokinetic parameter
Systemic Clearance From Plasma Following Extravascular Administration (CL/F) | From pre-dose on day 1 of cycle 1 to day 5 of cycle 3 (28-day cycle length)
  Pharmacokinetic parameter
The volume of distribution(Vd/F) | From pre-dose on day 1 of cycle 1 to day 5 of cycle 3 (28-day cycle length)
  Pharmacokinetic parameter
Average concentration at steady state(Cavg,ss) | From pre-dose on day 1 of cycle 1 to day 5 of cycle 3 (28-day cycle length)
  Pharmacokinetic parameter
Minimum observed concentration at steady state(Cmin,ss) | From pre-dose on day 1 of cycle 1 to day 5 of cycle 3 (28-day cycle length)
  Pharmacokinetic parameter

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No